CLINICAL TRIAL: NCT06377345
Title: Remote Patient Monitoring Solution for Chronic Respiratory Disease Management
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SingHealth Polyclinics (Other)
Responsible Party: Principal Investigator, Mabel Leow Qi He, Principle Investigator, SingHealth Polyclinics
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 202312-00011
Record Dates: First submitted 2024-04-08; First posted 2024-04-22 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Asthma; Asthma Attack; Asthma in Children; Asthma Acute; Asthma Chronic
MeSH Terms: conditions — Asthma | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: A two-group randomized controlled trial (RCT) design will be used. The control group will receive the usual care, and the intervention group will receive the Aevice device on top of usual care. Outcomes will be measured at baseline, week 4, and week 12. This is to evaluate the long-term impacts of the Aevice device. Clinicians who have interacted with participants using Aevice will also be invited to participate in an interview and clinician perception survey. A convenience sampling will be used for the recruitment of clinicians.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will not be aware of the participants' group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): The control group will receive the standard care provided by the Polyclinic. This can include a telephone follow-up by a nurse within 5 days, and follow-ups with a doctor after one week. All patients with asthma should also have an asthma action plan which provides them instructions on how to manage their asthma and the medications required when they experience symptoms. These symptoms include wheezing, chest tightness, difficulty breathing, coughing, night-waking, and symptom interfering with day-to-day activities.
  Interventions: Behavioral: Standard care
- Intervention group (Experimental): The intervention group will receive the AeviceMD device on top of standard care provided by the Polyclinic. They will use the AeviceMD device for 12 weeks. They are expected to use the device for at least 5 hours at night when they are asleep. However, they can also use the device at any time of the time, based on their own preference. The AeviceMD device will provide patients with objective information of their breathing (respiratory rate) and lung sounds. This objective information can be used for participants to self-manage their asthma following the asthma action plan. During the clinical follow-up, participants can show the clinician their lung parameters, to improve clinical management
  Interventions: Device: AeviceMD device; Behavioral: Standard care

INTERVENTIONS:
Device: AeviceMD device — The intervention group will receive the AeviceMD device on top of standard care provided by the Polyclinic. They will use the AeviceMD device for 12 weeks. They are expected to use the device for at least 5 hours at night when they are asleep. However, they can also use the device at any time of the time, based on their own preference. The AeviceMD device will provide patients with objective information of their breathing (respiratory rate) and lung sounds. This objective information can be used for participants to self-manage their asthma following the asthma action plan. During the clinical follow-up, participants can show the clinician their lung parameters, to improve clinical management
  Arms: Intervention group
Behavioral: Standard care — All participants will receive the standard care provided by the Polyclinic. This can include a telephone follow-up by a nurse within 5 days, and follow-ups with a doctor after one week. All patients with asthma should also have an asthma action plan which provides them instructions on how to manage their asthma and the medications required when they experience symptoms. These symptoms include wheezing, chest tightness, difficulty breathing, coughing, night-waking, and symptom interfering with day-to-day activities.

SUMMARY:
Aim: To evaluate the use of AeviceMD Monitoring System (AeviceMD) asthma in reducing acute exacerbation.

Methodology: Using a randomized controlled trial design, this project aims evaluate the effectiveness of AeviceMD in improving patients' outcomes in terms of reducing exacerbation, healthcare utilization, improving quality of life, self-efficacy, and cost effectiveness. Paediatric patients above age 7 and adults will be recruited. The data follow-up period is 3 months. It will also evaluate the usability of the device from both patients' and clinicians' perspective. 180 patients (124 adults, 56 pediatrics) and 120 clinicians will be recruited.

Importance of study: This study will evaluate if the AeviceMD can help improve disease management and reduce recurrence of asthma exacerbation.

Potential benefits and risk: AeviceMD allows for remote monitoring and tracking of patients' lung sounds, which could be used by patients to monitor their lung condition and prevent an episode of exacerbation or worsening exacerbations culminating in an admission which who further utilize already limited healthcare resources. An exacerbation is an episode of severe shortness of breath, cough, and chest tightening which warrants a visit to a healthcare institution. Through self-monitoring, patients can be empowered to self-manage their asthma, with aid of the asthma action plan which is given to all patients with asthma. AeviceMD can also help provide clinicians with patients' objective lung data. In the primary care setting, care is also fragmented as patients are often followed-up by a different doctor or healthcare providers. Clinicians have no objective data to track patients, and is dependent on patients' self-report and possible recall bias. There is no expected risk with the use of the device.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the clinical outcomes, self-efficacy, quality of life, utility, and cost-effectiveness of the Aevice device for asthma self-management post exacerbation.

The objectives are to evaluate:

1. The impact of Aevice on asthma symptom control (using Global Initiative for Asthma (GINA) score)
2. The impact of Aevice on asthma exacerbation (measure by number of rescue therapy, dose of oral Prednisolone used, referral to emergency department, and hospitalization)
3. The impact of Aevice on quality of life (using Euro Quality of Life - 5 Dimensions (E!Q5D) and mini-asthma quality of life questionnaire)
4. The patients' self-efficacy using Aevice (self-developed questionnaire)
5. The usability (system usability scale) and utility of Aevice (time of use and frequency of use)
6. The take-up rate and demographics of participants who accept versus decline the use of Aevice
7. Amount patients are willing to pay for the use of Aevice
8. Clinician perception and acceptability of using technology for telemonitoring and Aevice device
9. Evaluate the cost effectiveness of using Aevice

The ratio of adults to pediatrics exacerbation based on our statistics is 10:3 currently. To eliminate bias in age during randomization, stratified sampling is adopted, with a proposed mix of 126 adults and 54 pediatrics (63 adults and 27 pediatrics in each group).

Patients in each of the strata will be randomized in a 1:1 ratio to either intervention or control group according to a computer generated block randomization list. Random permuted blocks are used to ensure balance over time. The block size is determined by the study statistician and will kept confidential from the study team until final database lock. Each Patient will be assigned an individual randomization number upon randomization. This randomization number assigned will identify the patient and will be used for all documentation for this patient in this study. After the patient is screened eligibility and consented to the study, the site coordinator will call the centralized team for the randomization number and assignment. Blinding is not possible in the study team and patient as the intervention group will be receiving the new device.

Control group

The control group will receive the standard care provided by the Polyclinic. This can include a telephone follow-up by a nurse within 5 days, and follow-ups with a doctor after one week. All patients with asthma should also have an asthma action plan which provides them instructions on how to manage their asthma and the medications required when they experience symptoms. These symptoms include wheezing, chest tightness, difficulty breathing, coughing, night-waking, and symptom interfering with day-to-day activities.

Intervention

The intervention group will receive the Aevice device on top of standard care provided by the Polyclinic. They will use the Aevice device for 12 weeks. They are expected to use the device for at least 5 hours at night when they are asleep. However, they can also use the device at any time of the time, based on their own preference. The Aevice device will provide patients with objective information of their breathing (respiratory rate) and lung sounds. This objective information can be used for participants to self-manage their asthma following the asthma action plan. During the clinical follow-up, participants can show the clinician the their lung data from the Aevice application on their phone, for the clinician

The research coordinator will provide the participants with the Aevice device, and download the application on the participants' phone. The participant will be able to observe their trend on the application's dashboard They will be informed to share their lung parameters with their nurse during the follow-up call, and show the doctor data on their lung sounds during the follow-up visit. Participants will return the device at the end of the study period.

The participants will be instructed to contact the research coordinator if they face difficulties using the device. This will include problems with the Aevice device and phone application, or participants' do not know how to use the application.

Recruitment

Rescue therapy is administered by the nurses. The nurses in the Polyclinics will help identify patients in the treatment room who meet the inclusion criteria, and invite them to participate in the study. If the patient is agreeable, the nurse will refer the potential participant to the research coordinator. The doctors who are attending to patients with asthma exacerbation can also refer the patient to the research coordinator. The research coordinator will provide the participant information sheet (PIS), explain the details of the study, and go through the consent process with the participant. If the potential participant agrees to participate in the study, written informed consent will be obtained. After obtaining the informed consent, the research coordinator will collect the baseline data from the participant, allocate them to the group, and provide participants in the intervention group with the device.

The clinicians will be invited by email to participate in the survey and qualitative interview study, with a participant information sheet to understand the study rationale. If they agree to participate, the survey will be sent to them. They can participate in the survey only, and not the qualitative interview.

This study will be conducted at SingHealth Polyclinics.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma
* Pediatric patients (age 7 to 17), adult patients (age 18 and above
* Have an asthma exacerbation on the day of visit
* Be willing to use the AeviceMD device
* Has a smart phone to download the application that is paired with Aevice
* Has wireless fidelity (WIFI) connection to use with Aevice
* English speaking

Exclusion Criteria:

* No capacity for consent
* Concurrent chronic obstructive pulmonary disease (COPD)

Ages: 7 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Rescue therapy | up to 12 weeks
  number of times
Dose of oral Prednisolone use | up to 12 weeks
  Total dose in mg
Visit to hospital emergency department | up to 12 weeks
  number of times
Hospitalisation | up to 12 weeks
  total number of days
Euro Quality of Life 5 dimensions (EQ5D) | up to 12 weeks (baseline, week 4, week, 12)
  The Euro Quality of Life 5 dimension evaluates five items related to health: 1. mobility, 2. self-care, 3. usual activities, 4. pain/discomfort, and 5. anxiety/depression. A 5-point Likert scale is used for adults, ranging from no problems, slight problems, moderate problems, severe problems, and extreme problems. Scores from the five items can be used to derive a single utility score.
Asthma quality of life questionnaire (AQLQ) | up to 12 weeks (baseline, week 4, week, 12)
  The asthma quality of life questionnaire (AQLQ) will be used for participants above age 18. It consists of 32 items divided into four sections: symptoms (11 items), activity limitations (12 items), emotional function (5 items), and environmental stimuli (4 items). The intraclass correlation coefficient is 0.95. Each question is rated on a 7-point Likert scale. The Cronbach alpha is 0.9.
Pediatric asthma quality of life questionnaire (PAQLQ) | up to 12 weeks (baseline, week 4, week, 12)
  The Paediatric asthma quality of life questionnaire (PAQLQ) will be used for Paediatrics age 7 to 17. It consists of 23 items in 3 domains: activity limitation (5 items), symptoms (10 items) and emotional function (8 items). The questionnaire has been validated in Singapore, with intraclass correlation coefficient of 0.71

SECONDARY OUTCOMES:
Self-efficacy | up to 12 weeks, intervention group
  Self-efficacy will be measured using a self-developed questionnaire consisting of 6 questions. Each question will be rated on a 5-point Likert scale (strongly agree to strongly disagree). This is to evaluate if Aevice was useful for self-management of asthma
Usability | up to 12 weeks, intervention group
  The usability of device will be measured using the system usability scale (SUS). The scale consists of 10 items, rated on a 5-point Likert scale (score 1 to 5), with scores ranging from 10 to 50. Higher scores represent higher usability.
Heart rate | Throughout 12 weeks of study, intervention group
  Heart rate per minute, data obtained from the device. to record the average heart rate, and frequency of being out of range.
Respiratory rate | Throughout 12 weeks of study, intervention group
  respiratory rate per minute, data obtained from the device. To track average respiratory rate, and frequency of being out of range
Wheeze detection trend | Throughout 12 weeks of study, intervention group
  wheeze detection, data obtained from the device. The number of wheeze per day, and number of days with wheeze will be recorded
Medication log | Throughout 12 weeks of study, intervention group
  participant self entry of medication into the application, which will be obtained from the application. This will track patient frequency of taking inhaler
Duration of device usage | Throughout 12 weeks of study, intervention group
  number of hours use per day on average, and number of days used
Payment | 12 week, intervention group
  Amount the patient is willing to pay for the use of the device, in Singapore dollars

CONTACTS AND LOCATIONS:
Overall Officials: Mabel QH Leow, PhD, Principal Investigator — SingHealth Polyclinics
Locations (1):
- SingHealth Polyclinics, Singapore, Singapore